CLINICAL TRIAL: NCT05301010
Title: Randomized, Single-blind, Multicenter, Parallel Group Clinical Trial to Assess Efficacy and Safety of NNG-TMAB (Trastuzumab) in Combination With Docetaxel on Recurrent or Metastatic Breast Cancer Patients With Positive HER2
Brief Title: Clinical Trial to Assess Efficacy and Safety of NNG-TMAB (Trastuzumab) on Recurrent or Metastatic Breast Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nanogen Pharmaceutical Biotechnology Joint Stock Company (Industry)
Collaborators: Vietstar Biomedical Research (Industry); MedProve Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NNG17.2
Record Dates: First submitted 2022-03-17; First posted 2022-03-29 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer Metastatic; Breast Cancer Recurrent; Breast Cancer Female
MeSH Terms: interventions — Trastuzumab; Docetaxel

STUDY DESIGN:
Intervention Model Description: Two group: study drug and reference
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Faceptor + Docetacel (Experimental): Patients received a loading dose of Faceptor 8 mg/kg IV + docetaxel 75 mg/m^2 IV on Cycle 1 followed by Faceptor 6 mg/kg IV + docetaxel 75 mg/m^2 IV on the next 5 cycles (each cycle is 21 days)
  Interventions: Drug: Faceptor; Drug: Docetaxel
- Herceptin + Docetacel (Active Comparator): Patients received a loading dose of Herceptin 8 mg/kg IV + docetaxel 75 mg/m^2 IV on Cycle 1 followed by Herceptin 6 mg/kg IV + docetaxel 75 mg/m^2 IV on the next 5 cycles (each cycle is 21 days)
  Interventions: Drug: Herceptin; Drug: Docetaxel

INTERVENTIONS:
Drug: Faceptor — NNG-TMAB (trastuzumab) 150 mg, 440 mg, lyophilized power for injection, manufacturered by Nanogen Pharmaceutical Biotechnology JSC.
  Other Names: NNG-TMAB; Trastazumab
  Arms: Faceptor + Docetacel
Drug: Herceptin — Herceptin (trastuzumab) 150mg, 440mg, powder for concentrate for solution, manufactured by Roche.
  Other Names: Trastazumab
  Arms: Herceptin + Docetacel
Drug: Docetaxel — The drug Docetaxel in this study has the brand name Taxotere manufactured by Sanofi company.
  Other Names: Taxotere

SUMMARY:
Targeted therapy in the treatment of breast cancer targets HER2 receptor (Human Epidermal growth factor Receptor). HER2 receptor plays an important role in cell growth and differentiation (5). However, when HER2 overexpresses, it may lead to cancer. HER2 positive malignance exacerbates pathology and worsens clinical outcome, such as shortened overall survival (OS) compared with non-HER2 overexpression patients (6), (7). About 20-30% overexpression HER2/neogene breast cancer patients and patients having HER2 overexpression tumor have disease progression and poor prognosis in metastatic process (8), (9).

Currently, targeted therapeutic, which attaches to the HER2 receptor, inhibiting the growth of cancer cells has been approved. One of these products is Trastuzumab.

The study processed on 128 females aged between 18 and 65, recurrent or metastatic breast cancer patients with positive HER2.

The subjects were randomly distributed in 2 groups as NNG-TMAB + docetaxel or Herceptin® + docetaxel, in blocks of 4 in a 1: 1 ratio (NNG-TMAB: Herceptin®). In each block of 4 will be 2 patients in the experimental group and 2 patients in the control group

Primany endpoints is Overall Response Rate (ORR) according to RECIST 1.1. ORR includes Complete Response Rate and Partial Response Rate. ORR will be independently evaluated by an Independent Tumor Evaluation Board (ITEB).

This trial is intended to assess the biosimilarity of efficacy and safety between NNG-TMAB (Trastuzumab) and Herceptin® in combination with Docetaxel on recurrent or metastatic breast cancer patients with positive HER2.

ELIGIBILITY:
Inclusion Criteria:

* Female patients from 18 to 65 years old.
* Willing to give written and signed informed consent.
* Have pathologically or cytologically confirmed breast cancer.
* Inoperable, recurrent or metastatic breast cancer according to TNM classification and investigator' s assessment.
* Presence of at least 1 tumour with a size not less than 1 cm (revealed with computed tomography (CT) slice thickness not more than 5 mm). Patients having bone metastasis as the only measurable tumour are not eligible for the trial.
* Grade 3+ HER2 overexpression confirmed by immunohistochemical (IHC) staining or grade 2+ HER2 overexpression accompanied by HER2 gene amplification confirmed by fluorescent hybridization in situ (FISH).
* Eastern Cooperative oncology group performance status ≤ 2
* Willing to comply the requirements of the study protocol.
* Have a survival expectancy of at least 6 months.
* At screening period: Hb ≥ 9 g/dL; Neutrophils ≥ 1,5x10^9/L; platelets ≥ 100x10^9/L; creatinine level ≤ 1,5 x upper limit of normal (ULN); bilirubin level < 1,5 x ULN; ALT/AST < 2,5 x ULN (< 5 x ULN for patients with liver metastases), ALP < 5 x ULN.
* Patients of childbearing potential and her partner must implement reliable contraceptive measures during the study treatment, starting 4 weeks prior to inclusion into the trial and until 6 months after the last administration of the study drug

Exclusion Criteria:

* Previous anticancer therapy for metastatic BC, including previous anticancer therapy with signal transduction inhibitors (e.g. lapatinib), biological drugs (e.g. trastuzumab, bevacizumab), experimental (not approved for BC therapy) anticancer drugs. Any previous chemotherapy or hormonal therapy is allowed.
* Previously treated with doxorubicin > 400 mg/m2; epirubicin > 800 mg/m2 in accumulative dosages.
* Surgery, radiation therapy, use of any experimental medications within 4 weeks prior to randomization.
* Clinical evidence or X-ray show that breast cancer metastases in central nervous system
* Patients with metastatic tumor to the bone is the only tumor to be measured
* Systolic blood pressure >150mmHg and/or diastolic blood pressure >100mmHg. Uncontrolled hypertension comprising all cases of arterial hypertension when no decrease in blood pressure could be achieved despite treatment with a combination of 3 antihypertensive drugs including one diuretic and non-medicamental correction methods (low salt diet, physical exercise)
* Cardiovascular system pathology (congestive heart failure (CHF) stage III-IV according to New York Heart Association (NYHA) classification, unstable angina pectoris, myocardial infarction) within 12 months prior to randomization. LVEF < 50% according to echocardiogram when screening.
* Acute or chronic infection (except for acute or chronic infection that is stable and does not affect the study evaluation). Infecting HIV, HBV or HCV, Syphilis
* Patients with a history of severe allergic reaction to trastuzumab, paclitaxel, docetaxel or other ingredients in the formulation
* The patient has evidence of a serious illness (such as resting dyspnea or severe lung disease, etc.) or an abnormal laboratory test that, in the judgment of the researcher, will affect participation. research and completion of patient research, or may affect the patient's response evaluation.
* Pregnancy, intend to get pregnant, lactation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) according to RECIST 1.1 after 6 cycles | at the end of cycle 6 (each cycle is 21 days)
  ORR includes Complete Response Rate and Partial Response Rate. ORR will be independently evaluated by an Independent Tumor Evaluation Board (ITEB).
Overall Response Rate (ORR) according to RECIST 1.1 at the end of study | baseline through end of study (up to 128 days)
  ORR includes Complete Response Rate and Partial Response Rate. ORR will be independently evaluated by an Independent Tumor Evaluation Board (ITEB).

SECONDARY OUTCOMES:
Progressive Disease Rate (PDR) according to RECIST 1.1 | PDR will be evaluated every 3 cycles (each cycle is 21 days) through the end of study (up to 128 days)
  Progressive Disease Rate (PDR). PDR will be independently evaluated by an Independent Tumor Evaluation Board (ITEB).
Stable Disease Rate (SDR) according to RECIST 1.1 | SDR will be evaluated every 3 cycles (each cycle is 21 days) through the end of study (up to 128 days)
  Stable Disease Rate (SDR). SDR will be independently evaluated by an Independent Tumor Evaluation Board (ITEB).
Progression-free survival (PFS) according to RECIST 1.1 | Baseline up to disease progression or death due to any cause, whichever occurs first (up to 128 days (6 cycles - each cycle is 21 days))
  Progression-free survival (PFS) was defined as the time between the date patient signed the Informed Consent Form (ICF) and the date of disease progression or death from any cause.
Evaluate the patient's quality of life | At week 24th
  Quality of life of patients according to the EORTC QLQ-C30 questionnaire combined with EORTC QLQ-BR23 at week 24. All scores were linearly transformed to a 0 to 100 scale, according to international guidelines before assessment. A high or healthy level of functioning is represented by a high functional score. A high QOL is represented by a high score for global health status or QOL. More severe symptoms or problems are represented by high symptom scores or items.
  (i) EORTC QLQ-C30: is designed to measure cancer patients' physical, psychological and social functions.
  (ii) EORTC QLQ-BR23: is a breast-specific module that comprises of 23 questions.
Anti-drug antibody evaluation | At baseline,after 3 cycles of treatment, after 6 cycles of treatment (each cycle is 21 days)
  Percentage of participants with positive Anti-drug antibody
Rate of AE and SAE occurence | up to 128 days (6 cycles - each cycle is 21 days)
  Frequency of adverse events, including clinical examination, vital signs and laboratory tests

CONTACTS AND LOCATIONS:
Locations (2):
- Vietnam (2):
  - 19-8 Hospital, Hanoi
  - HCMC Oncology Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bullock K, Blackwell K. Clinical efficacy of taxane-trastuzumab combination regimens for HER-2-positive metastatic breast cancer. Oncologist. 2008 May;13(5):515-25. doi: 10.1634/theoncologist.2007-0204. PMID 18515736
- [Background] Polychemotherapy for early breast cancer: an overview of the randomised trials. Early Breast Cancer Trialists' Collaborative Group. Lancet. 1998 Sep 19;352(9132):930-42. PMID 9752815
- [Background] Gennari A, Conte P, Rosso R, Orlandini C, Bruzzi P. Survival of metastatic breast carcinoma patients over a 20-year period: a retrospective analysis based on individual patient data from six consecutive studies. Cancer. 2005 Oct 15;104(8):1742-50. doi: 10.1002/cncr.21359. PMID 16149088
- [Background] Hynes NE, Stern DF. The biology of erbB-2/neu/HER-2 and its role in cancer. Biochim Biophys Acta. 1994 Dec 30;1198(2-3):165-84. doi: 10.1016/0304-419x(94)90012-4. No abstract available. PMID 7819273
- [Background] Slamon DJ, Clark GM, Wong SG, Levin WJ, Ullrich A, McGuire WL. Human breast cancer: correlation of relapse and survival with amplification of the HER-2/neu oncogene. Science. 1987 Jan 9;235(4785):177-82. doi: 10.1126/science.3798106.
- [Background] Slamon DJ, Godolphin W, Jones LA, Holt JA, Wong SG, Keith DE, Levin WJ, Stuart SG, Udove J, Ullrich A, et al. Studies of the HER-2/neu proto-oncogene in human breast and ovarian cancer. Science. 1989 May 12;244(4905):707-12. doi: 10.1126/science.2470152.
- [Background] Press MF, Bernstein L, Thomas PA, Meisner LF, Zhou JY, Ma Y, Hung G, Robinson RA, Harris C, El-Naggar A, Slamon DJ, Phillips RN, Ross JS, Wolman SR, Flom KJ. HER-2/neu gene amplification characterized by fluorescence in situ hybridization: poor prognosis in node-negative breast carcinomas. J Clin Oncol. 1997 Aug;15(8):2894-904. doi: 10.1200/JCO.1997.15.8.2894. PMID 9256133
- [Background] Marty M, Cognetti F, Maraninchi D, Snyder R, Mauriac L, Tubiana-Hulin M, Chan S, Grimes D, Anton A, Lluch A, Kennedy J, O'Byrne K, Conte P, Green M, Ward C, Mayne K, Extra JM. Randomized phase II trial of the efficacy and safety of trastuzumab combined with docetaxel in patients with human epidermal growth factor receptor 2-positive metastatic breast cancer administered as first-line treatment: the M77001 study group. J Clin Oncol. 2005 Jul 1;23(19):4265-74. doi: 10.1200/JCO.2005.04.173. Epub 2005 May 23. PMID 15911866
- [Background] Ahuja SP, Mehta SK. Incorporation of 2-14C-acetate into the lipids of various membranes from buffalo milk. Zentralbl Veterinarmed A. 1979 May;26(4):318-26. doi: 10.1111/j.1439-0442.1979.tb01762.x. No abstract available. PMID 113962
- [Background] Plosker GL, Keam SJ. Trastuzumab: a review of its use in the management of HER2-positive metastatic and early-stage breast cancer. Drugs. 2006;66(4):449-75. doi: 10.2165/00003495-200666040-00005. PMID 16597163
- [Background] Meza-Junco J, Au HJ, Sawyer MB. Trastuzumab for gastric cancer. Expert Opin Biol Ther. 2009 Dec;9(12):1543-51. doi: 10.1517/14712590903439702. PMID 19916733
- [Background] Lara PN Jr, Chee KG, Longmate J, Ruel C, Meyers FJ, Gray CR, Edwards RG, Gumerlock PH, Twardowski P, Doroshow JH, Gandara DR. Trastuzumab plus docetaxel in HER-2/neu-positive prostate carcinoma: final results from the California Cancer Consortium Screening and Phase II Trial. Cancer. 2004 May 15;100(10):2125-31. doi: 10.1002/cncr.20228. PMID 15139054
- [Background] Tedesco KL, Thor AD, Johnson DH, Shyr Y, Blum KA, Goldstein LJ, Gradishar WJ, Nicholson BP, Merkel DE, Murrey D, Edgerton S, Sledge GW Jr. Docetaxel combined with trastuzumab is an active regimen in HER-2 3+ overexpressing and fluorescent in situ hybridization-positive metastatic breast cancer: a multi-institutional phase II trial. J Clin Oncol. 2004 Mar 15;22(6):1071-7. doi: 10.1200/JCO.2004.10.046. PMID 15020608
- [Background] [Study Results] Bines J, Murad A et al. (2003), Weekly docetaxel (Docetaxel) and trastuzumab (Herceptin) as primary therapy in stage III, HER2 overexpressing breast cancer - a Brazilian multicenter study. Breast cancer Res Treat, 82 (suppl 1):S56
- [Background] Pivot X, Romieu G, Debled M, Pierga JY, Kerbrat P, Bachelot T, Lortholary A, Espie M, Fumoleau P, Serin D, Jacquin JP, Jouannaud C, Rios M, Abadie-Lacourtoisie S, Tubiana-Mathieu N, Cany L, Catala S, Khayat D, Pauporte I, Kramar A; PHARE trial investigators. 6 months versus 12 months of adjuvant trastuzumab for patients with HER2-positive early breast cancer (PHARE): a randomised phase 3 trial. Lancet Oncol. 2013 Jul;14(8):741-8. doi: 10.1016/S1470-2045(13)70225-0. Epub 2013 Jun 11. PMID 23764181
- [Background] Wardley AM, Pivot X, Morales-Vasquez F, Zetina LM, de Fatima Dias Gaui M, Reyes DO, Jassem J, Barton C, Button P, Hersberger V, Torres AA. Randomized phase II trial of first-line trastuzumab plus docetaxel and capecitabine compared with trastuzumab plus docetaxel in HER2-positive metastatic breast cancer. J Clin Oncol. 2010 Feb 20;28(6):976-83. doi: 10.1200/JCO.2008.21.6531. Epub 2009 Dec 28. PMID 20038734
- [Background] Bell R. What can we learn from Herceptin trials in metastatic breast cancer? Oncology. 2002;63 Suppl 1:39-46. doi: 10.1159/000066200. PMID 12422054
- [Background] Harvey V, Mouridsen H, Semiglazov V, Jakobsen E, Voznyi E, Robinson BA, Groult V, Murawsky M, Cold S. Phase III trial comparing three doses of docetaxel for second-line treatment of advanced breast cancer. J Clin Oncol. 2006 Nov 1;24(31):4963-70. doi: 10.1200/JCO.2005.05.0294. Epub 2006 Oct 10. PMID 17033039
- [Background] Chan S, Friedrichs K, Noel D, Pinter T, Van Belle S, Vorobiof D, Duarte R, Gil Gil M, Bodrogi I, Murray E, Yelle L, von Minckwitz G, Korec S, Simmonds P, Buzzi F, Gonzalez Mancha R, Richardson G, Walpole E, Ronzoni M, Murawsky M, Alakl M, Riva A, Crown J; 303 Study Group. Prospective randomized trial of docetaxel versus doxorubicin in patients with metastatic breast cancer. J Clin Oncol. 1999 Aug;17(8):2341-54. doi: 10.1200/JCO.1999.17.8.2341. PMID 10561296
- [Background] Joensuu H, Bono P, Kataja V, Alanko T, Kokko R, Asola R, Utriainen T, Turpeenniemi-Hujanen T, Jyrkkio S, Moykkynen K, Helle L, Ingalsuo S, Pajunen M, Huusko M, Salminen T, Auvinen P, Leinonen H, Leinonen M, Isola J, Kellokumpu-Lehtinen PL. Fluorouracil, epirubicin, and cyclophosphamide with either docetaxel or vinorelbine, with or without trastuzumab, as adjuvant treatments of breast cancer: final results of the FinHer Trial. J Clin Oncol. 2009 Dec 1;27(34):5685-92. doi: 10.1200/JCO.2008.21.4577. Epub 2009 Nov 2. PMID 19884557
- [Background] Baselga J, Carbonell X, Castaneda-Soto NJ, Clemens M, Green M, Harvey V, Morales S, Barton C, Ghahramani P. Phase II study of efficacy, safety, and pharmacokinetics of trastuzumab monotherapy administered on a 3-weekly schedule. J Clin Oncol. 2005 Apr 1;23(10):2162-71. doi: 10.1200/JCO.2005.01.014. PMID 15800309
- [Background] Hamberg P, Bos MM, Braun HJ, Stouthard JM, van Deijk GA, Erdkamp FL, van der Stelt-Frissen IN, Bontenbal M, Creemers GJ, Portielje JE, Pruijt JF, Loosveld OJ, Smit WM, Muller EW, Schmitz PI, Seynaeve C, Klijn JG; Dutch Breast Cancer Trialists' Group (BOOG). Randomized phase II study comparing efficacy and safety of combination-therapy trastuzumab and docetaxel vs. sequential therapy of trastuzumab followed by docetaxel alone at progression as first-line chemotherapy in patients with HER2+ metastatic breast cancer: HERTAX trial. Clin Breast Cancer. 2011 Apr;11(2):103-13. doi: 10.1016/j.clbc.2011.03.003. Epub 2011 Apr 11. PMID 21569996